CLINICAL TRIAL: NCT02265237
Title: A Randomized, Open-Label Study to Evaluate the Safety and Efficacy of Ombitasvir/ABT-450/Ritonavir Co-administered With Ribavirin (RBV) in Adults With Genotype 4 Chronic Hepatitis C Virus (HCV) Infection and Cirrhosis (AGATE-1)
Acronym: AGATE-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M11-665; 2014-001496-31 (EudraCT Number)
Record Dates: First submitted 2014-10-10; First posted 2014-10-15 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Hepatitis C Virus
Keywords: Compensated Cirrhosis; Hepatitis C; Hepatitis C Genotype 4; Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — ombitasvir; Ritonavir; paritaprevir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A (Experimental): Ombitasvir/paritaprevir/ritonavir (25/150/100 mg) and Ribavirin dosed for 12 weeks for genotype 4 treatment-naïve or treatment-experienced with IFN/RBV.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir; Drug: ribavirin
- Arm B (Experimental): Ombitasvir/paritaprevir/ritonavir (25/150/100 mg) and Ribavirin dosed for 16 weeks for genotype 4 treatment-naive or treatment-experienced with IFN/RBV.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir; Drug: ribavirin
- Arm C (Experimental): Ombitasvir/paritaprevir/ritonavir (25/150/100 mg) and Ribavirin dosed for 24 weeks for genotype 4 treatment-naive and treatment-experienced with IFN/RBV.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir; Drug: ribavirin
- Arm D (Experimental): Ombitasvir/paritaprevir/ritonavir (25/150/100 mg) and Ribavirin dosed for 24 weeks for genotype 4 SOF/pegIFN/RBV or SOF/RBV treatment-experienced.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir; Drug: ribavirin

INTERVENTIONS:
Drug: ombitasvir/paritaprevir/ritonavir — tablets
  Other Names: norvir (ritonavir); paritaprevir (ABT-450); ombitasvir (ABT-267)
Drug: ribavirin — tablets

SUMMARY:
The purpose of this study in HCV genotype 4-infected participants with compensated cirrhosis is to assess the safety and to compare the percentage of participants achieving a 12-week sustained virologic response (SVR12), [HCV ribonucleic acid (RNA) < lower limit of quantification (LLOQ) 12 weeks following treatment], to a clinically relevant threshold [based on SVR rates for HCV genotype 4-infected participants treated with pegylated interferon (pegIFN)/RBV].

DETAILED DESCRIPTION:
This is a Phase 3, randomized, open-label, multicenter study evaluating the safety and efficacy of ombitasvir/paritaprevir/ritonavir coadministered with RBV for 12, 16, or 24 weeks in HCV genotype 4 (GT4)-infected participants with compensated cirrhosis who are either treatment-naïve or who had previously received only IFN/RBV treatment for HCV.

The study also enrolled HCV GT4-infected participants with compensated cirrhosis who had previously experienced virologic failure with either SOF/pegIFN/RBV or sofosbuvir (SOF)/RBV treatment. These participants were treated with ombitasvir/paritaprevir/ritonavir coadministered with RBV for 24 weeks in this study.

This study was divided into 2 parts with approximately 184 total participants. Part I included participants who were randomized to receive either 12 or 16 weeks of treatment and Part II included participants who received 24 weeks of treatment. Enrollment into Part II opened once randomization in Part I was completed.

ELIGIBILITY:
Inclusion Criteria:

For Arms A, B and C:

- Participants must meet one of the following:

* Treatment-naive: Participant has never received antiviral treatment for hepatitis C infection OR
* Treatment Experienced (Prior null responders, Partial responders or Relapsers to IFN/RBV);

For Arm D:

- Participant must have prior treatment experience with SOF/pegIFN/RBV or SOF/RBV and meet one of the following categories:

* Prior SOF breakthrough/non-responder: HCV RNA detectable at the end of treatment with SOF/pegIFN/RBV or SOF/RBV;
* Prior SOF relapser: achieved HCV RNA undetectable at end of a prior treatment course SOF/pegIFN/RBV or SOF/RBV, but HCV RNA was detectable within 52 weeks following completion of therapy.

For Arms A, B, C and D:

* Chronic HCV genotype 4 infection with cirrhosis.
* Participant has plasma HCV RNA level > 1,000 IU/mL at Screening

Exclusion Criteria:

* Positive test result at Screening for Hepatitis B surface antigen (HBsAg) or anti-human immunodeficiency virus antibody (HIV Ab).
* Current enrollment in another interventional clinical study, previous enrollment in this study, or previous use of any protease inhibitor, non-nucleoside polymerase inhibitor, or Nonstructural viral protein (NS) 5A inhibitor, either investigational or commercially available (including previous exposure to paritaprevir or ombitasvir), or receipt of any investigational product within 6 weeks prior to study drug administration. Prior use of any direct-acting antiviral will not be allowed, except for Arm D where prior experience with the nucleoside polymerase inhibitor, sofosbuvir with pegIFN/RBV or SOF with RBV is required.
* Any current or past clinical evidence of Child-Pugh B or C classification or clinical history of liver decompensation including ascites, variceal bleeding, or hepatic encephalopathy.
* Confirmed presence of hepatocellular carcinoma.
* Any cause of liver disease other than chronic HCV infection.
* Abnormal laboratory tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2014-10-28; Primary Completion 2016-07-28 (Actual); Study Completion 2017-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

REFERENCES:
- [Derived] Asselah T, Hezode C, Qaqish RB, ElKhashab M, Hassanein T, Papatheodoridis G, Feld JJ, Moreno C, Zeuzem S, Ferenci P, Yu Y, Redman R, Pilot-Matias T, Mobashery N. Ombitasvir, paritaprevir, and ritonavir plus ribavirin in adults with hepatitis C virus genotype 4 infection and cirrhosis (AGATE-I): a multicentre, phase 3, randomised open-label trial. Lancet Gastroenterol Hepatol. 2016 Sep;1(1):25-35. doi: 10.1016/S2468-1253(16)30001-2. Epub 2016 Jun 16. PMID 28404108

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was divided into 2 parts with 184 total participants. Part I (Arms A and B) included participants who received either 12 or 16 weeks of treatment and Part II (Arms C and D) included participants who received 24 weeks of treatment. Enrollment into Part II opened once randomization in Part I was completed.
Pre-assignment Details: Safety analysis population: all participants who received at least 1 dose of study drug. One participant randomized to the arm B (16 weeks arm) was erroneously administered study drug for 12 weeks (as in arm A). Therefore this participant is included in arm A for the safety population.
Period: As Enrolled (Overall Study)
Arm/Group | Arm A | Arm B | Arm C | Arm D
Started | 59 | 61 | 61 | 3
Completed | 54 | 58 | 51 | 2
Not Completed | 5 | 3 | 10 | 1
Period: As Treated (Overall Study)
Arm/Group | Arm A | Arm B | Arm C | Arm D
Started | 60 (One arm B subject received the drug for the duration for arm A and was included in arm A for safety.) | 60 (One arm B subject received the drug for the duration for arm A and was included in arm A for safety.) | 61 | 3
Completed | 55 | 57 | 51 | 2
Not Completed | 5 | 3 | 10 | 1
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 2 | 6 | 0
Not completed — Other | 2 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis population: all participants who received at least 1 dose of study drug. One participant randomized to arm B (16 weeks arm) was erroneously administered study drug for 12 weeks (as in arm A). Therefore this participant is included in arm A for the safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Arm D | Total
Number analyzed (Participants) | 60 | 60 | 61 | 3 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (8.08) | 57.1 (9.08) | 54.6 (9.02) | 62.3 (8.08) | 56.6 (8.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 22 | 18 | 0 | 54
  Male | 46 | 38 | 43 | 3 | 130
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 6 | 0 | 9
  Not Hispanic or Latino | 58 | 59 | 55 | 3 | 175
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Arms A, B and C With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification (<LLOQ) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug
Population: Intent-to-treat (ITT) population: all participants who received at least 1 dose of study drug; participants with missing data after backwards imputation were imputed as nonresponders.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 59 | 61 | 61
percentage of participants | 96.6 [86.7 to 99.2] | 100.0 [92.4 to 100.0] | 93.4 [82.6 to 97.7]
Statistical Analysis 1: Comparison: Arm B; The overall 2-sided significance level of 0.05 was split between Part I (arms A and B) and Part II (arm C) using a Bonferroni corrected alpha level of 0.025 for each part. Additionally, a fixed sequence procedure for Part I was used to proceed through the primary efficacy comparisons in the following order: 1) test of superiority of arm B and 2) test of superiority of arm A. The primary outcome within Arm C was tested with a Bonferroni-corrected Type 1 error rate of 0.025 for superiority; Test type: Superiority — 97.5% CI was calculated using the Wilson score method; the lower confidence bound for the percentage of participants with sustained virologic response at 12 weeks after treatment must exceed 67% to achieve superiority. The predefined threshold of 67% was based on historical SVR rates for HCV genotype 4 (GT4)-infected subjects treated with pegIFN/RBV; Percentage of Participants = 100, 97.5% CI 2-sided [92.4 to 100.0] — The confidence interval was calculated using the Wilson score method
Statistical Analysis 2: Comparison: Arm A; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — 97.5% confidence interval (CI) was calculated using the Wilson score method; the lower confidence bound for the percentage of participants with sustained virologic response at 12 weeks after treatment must exceed 67% to achieve superiority. The predefined threshold of 67% was based on historical SVR rates for HCV GT4-infected subjects treated with pegIFN/RBV; Percentage of Participants = 96.6, 97.5% CI 2-sided [86.7 to 99.2] — The confidence interval was calculated using the Wilson score method
Statistical Analysis 3: Comparison: Arm C; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Percentage of Participants = 93.4, 97.5% CI 2-sided [82.6 to 97.7] — The confidence interval was calculated using the Wilson score method

2. Secondary Outcome: Percentage of Participants With SVR12 in Participants Receiving 12 Weeks (Arm A) of Treatment Compared to Participants Receiving 16 Weeks of Treatment (Arm B)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug
Population: All participants who received at least 1 dose of study drug (ITT population); participants with missing data after backwards imputation were imputed as nonresponders.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 59 | 61
percentage of participants | 96.6 | 100
Statistical Analysis 1: Comparison: Arm A vs Arm B; Within Part I (arm A and B), since superiority was demonstrated for both arms in the primary outcome measures, testing continued to the first secondary outcome measure; Test type: Superiority — Treatment differences (with 95% confidence intervals) and corresponding P-value for the specified comparisons were estimated using stratum adjusted Mantel-Haenszel (MH) proportion and continuity-corrected variance, adjusting for IFN/RBV treatment history (treatment-naïve or treatment-experienced); p = 0.304, Mantel Haenszel; Stratum-Adjusted MH Difference = -3.39, 95% CI 2-sided [-9.85 to 3.07]

3. Secondary Outcome: Percentage of Participants With SVR12 in Participants Receiving 16 Weeks (Arm B) of Treatment Compared to Participants Receiving 24 Weeks of Treatment (Arm C)
Description: as for outcome 2
Time Frame: 12 weeks after the last actual dose of study drug
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Arm B | Arm C
Number analyzed (Participants) | 61 | 57
percentage of participants | 100 | 93.4
Statistical Analysis 1: Comparison: Arm B vs Arm C; Within Part II (arm C), since superiority was demonstrated for the primary outcome measure, testing continued to the second secondary outcome measure; Test type: Superiority — Treatment differences (with 95% confidence intervals) and corresponding P-value for the specified comparisons were estimated using stratum adjusted Mantel-Haenszel proportion and continuity-corrected variance, adjusting for IFN/RBV treatment history (treatment-naïve or treatment-experienced); p = 0.086, Mantel Haenszel; Stratum-Adjusted MH Difference = 6.45, 95% CI 2-sided [-0.91 to 13.81]

4. Secondary Outcome: Percentage of Participants in Arms A, B and C With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as confirmed HCV RNA ≥ LLOQ after HCV RNA < LLOQ during treatment; confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline in HCV RNA during treatment; or all on-treatment values of HCV RNA >= LLOQ with at least 6 weeks of treatment.
Time Frame: Up to Treatment Week 24 (end of treatment) or premature discontinuation from treatment
Population: All participants who received at least 1 dose of study drug (ITT population).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 59 | 61 | 61
percentage of participants | 1.7 [0.3 to 9.0] | 0 [0.0 to 5.9] | 0 [0.0 to 5.9]

5. Secondary Outcome: Percentage of Participants in Arms A, B and C With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants with HCV RNA levels < LLOQ at the end of treatment.
Time Frame: From the end of treatment through 12 weeks after the last dose of study drug
Population: All participants who received at least 1 dose of study drug (ITT population) with at least one post-treatment HCV RNA value, completed treatment, and had HCV RNA <LLOQ at the final treatment visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 57 | 59 | 56
percentage of participants | 0 [0.0 to 6.3] | 0 [0.0 to 6.1] | 0 [0.0 to 6.4]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration until 30 days after the last dose of study drug (up to 28 weeks)
Description: TEAEs and TESAEs are defined as any adverse event (AE) with an onset date that is after the first dose of study drug until 30 days after the last dose of study drug. TEAEs were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Arm A | Arm B | Arm C | Arm D
Serious Adverse Events (participants affected / at risk) | 4/60 | 4/60 | 3/61 | 0/3
Other Adverse Events (participants affected / at risk) | 46/60 | 55/60 | 50/61 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=60) | Arm B (N=60) | Arm C (N=61) | Arm D (N=3)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 2 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 1 | 0
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 0
HEPATOTOXICITY (Hepatobiliary disorders) | 0 | 0 | 1 | 0
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 0 | 1 | 0 | 0
CLOSTRIDIUM COLITIS (Infections and infestations) | 0 | 1 | 0 | 0
MENINGITIS (Infections and infestations) | 0 | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 1 | 0 | 0
PNEUMONIA KLEBSIELLA (Infections and infestations) | 0 | 1 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
SCIATICA (Nervous system disorders) | 0 | 1 | 0 | 0
MANIA (Psychiatric disorders) | 1 | 0 | 0 | 0
SUICIDAL IDEATION (Psychiatric disorders) | 0 | 0 | 1 | 0
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=60) | Arm B (N=60) | Arm C (N=61) | Arm D (N=3)
ANAEMIA (Blood and lymphatic system disorders) | 7 | 12 | 7 | 0
EAR PAIN (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 4 | 6 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 | 1 | 2 | 1
CONSTIPATION (Gastrointestinal disorders) | 4 | 1 | 2 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 3 | 2 | 0
NAUSEA (Gastrointestinal disorders) | 6 | 8 | 5 | 1
TOOTHACHE (Gastrointestinal disorders) | 2 | 3 | 2 | 0
VOMITING (Gastrointestinal disorders) | 4 | 3 | 4 | 0
ASTHENIA (General disorders) | 11 | 19 | 15 | 1
FATIGUE (General disorders) | 10 | 20 | 16 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 3 | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 5 | 4 | 2 | 0
PYREXIA (General disorders) | 0 | 3 | 1 | 0
JAUNDICE (Hepatobiliary disorders) | 3 | 2 | 4 | 0
SINUSITIS (Infections and infestations) | 0 | 3 | 0 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 1 | 3 | 0 | 0
HAEMOGLOBIN DECREASED (Investigations) | 3 | 8 | 4 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 5 | 2 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 4 | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 4 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 2 | 5 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 | 6 | 3 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 4 | 9 | 0 | 0
HEADACHE (Nervous system disorders) | 14 | 14 | 13 | 0
MEMORY IMPAIRMENT (Nervous system disorders) | 1 | 4 | 1 | 0
ANXIETY (Psychiatric disorders) | 3 | 2 | 3 | 0
INSOMNIA (Psychiatric disorders) | 5 | 6 | 5 | 1
SLEEP DISORDER (Psychiatric disorders) | 2 | 5 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 4 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 4 | 0
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
PARANASAL SINUS DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 1 | 4 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 5 | 14 | 12 | 1
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
RASH (Skin and subcutaneous tissue disorders) | 4 | 3 | 2 | 1
HYPERTENSION (Vascular disorders) | 4 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.